CLINICAL TRIAL: NCT00145470
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blinded Trial Evaluating the Safety and Efficacy of Asenapine in Subjects Continuing Lithium or Valproic Acid/Divalproex Sodium for the Treatment of an Acute Manic or Mixed Episode
Brief Title: 12 Week Study of the Safety/Efficacy of Asenapine When Added to Lithium/Valproate in the Treatment of Bipolar Disorder (A7501008 / P05844 / MK-8274-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05844; A7501008 (Other: Organon); 2004-003927-11 (EudraCT Number); MK-8274-017 (Other: Merck Protocol Number); P05844 (Other: Schering-Plough)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asenapine (Experimental): Participants received asenapine as a fast-dissolving sublingual (SL) tablet, given twice daily (BID). On Day 1, participants received asenapine 5 mg, BID. On Days 2 to 84, asenapine was dosed flexibly: BID at either 5 or 10 mg. Asenapine doses were up- or down-titrated based on efficacy, safety, and tolerability.
  Interventions: Drug: Asenapine
- Placebo (Placebo Comparator): Participants received placebo on Days 1-84 as a fast-dissolving SL tablet, BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — Asenapine fast dissolving SL tablets 5 and 10 mg; starting dose 5 mg BID on Day 1; 5-10 mg BID after Day 1.
  Other Names: Org 5222
  Arms: Asenapine
Drug: Placebo — Placebo fast dissolving SL tablets, BID
  Arms: Placebo

SUMMARY:
This is a 12-week study that will test the safety and efficacy of asenapine when used in addition to lithium or valproate for subjects with acute manic or mixed episodes of Bipolar I Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Have bipolar I disorder, current episode manic or mixed
* Treated with lithium or valproic acid

Exclusion Criteria:

* Have an unstable medical condition
* Clinically significant laboratory abnormality.
* Have a primary diagnosis other than bipolar I disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2005-06-02 (Actual); Primary Completion 2007-02-28 (Actual); Study Completion 2007-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szegedi A, Calabrese JR, Stet L, Mackle M, Zhao J, Panagides J; Apollo Study Group. Asenapine as adjunctive treatment for acute mania associated with bipolar disorder: results of a 12-week core study and 40-week extension. J Clin Psychopharmacol. 2012 Feb;32(1):46-55. doi: 10.1097/JCP.0b013e31823f872f. PMID 22198448

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo on Days 1-84 as a fast-dissolving sublingual (SL) tablet, given twice daily (BID).
- Asenapine: Participants received asenapine as a fast-dissolving SL tablet, BID. On Day 1, participants received asenapine 5 mg, BID. On Days 2 to 84, asenapine was dosed flexibly: BID at either 5 or 10 mg. Asenapine doses were up- or down-titrated based on efficacy, safety, and tolerability.
Period: Overall Study
Arm/Group | Placebo | Asenapine
Started | 167 | 159
Treated | 166 | 158
Completed | 55 | 61
Not Completed | 112 | 98
Not completed — Adverse Event | 19 | 25
Not completed — Lack of Efficacy | 27 | 13
Not completed — Withdrawal by Subject | 36 | 34
Not completed — Lost to Follow-up | 21 | 17
Not completed — Reason Not Reported | 9 | 9

BASELINE CHARACTERISTICS:
Population: Includes all participants receiving study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Asenapine | Total
Number analyzed (Participants) | 166 | 158 | 324
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (11.97) | 39.6 (11.71) | 39.3 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 137
  Male | 97 | 90 | 187

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in Young-Mania Rating Scale (Y-MRS) Score at Day 21
Description: The least squares mean change from baseline in Y-MRS score at day 21 was assessed. The Y-MRS is a clinician-rated instrument used for assessing the symptoms of mania, composed of 11 items. For the 11 items, scores range from 0 (symptoms absent) to, depending on the item, either 4 (7 items) or 8 (4 items). Scores for individual items add to a total score (range: 0-60), with higher scores indicating greater symptom severity. Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a last observation carried forward (LOCF) analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: Includes all randomized participants receiving ≥1 dose of study treatment, having ≥1 post-dose Y-MRS assessment.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline | 28.2 (0.45) | 27.9 (0.46)
  Change from Baseline at Day 21 | -7.9 (0.76) | -10.3 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.0257, ANCOVA — P-value based on the difference in the least squares (LS) means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

2. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: The number of participants experiencing an AE was assessed. An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the use of the investigational product, whether or not considered related to the investigational product.
Time Frame: Up to Day 114
Population: Includes all randomized participants receiving ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 166 | 158
Participants | 114 | 116

3. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: The number of participants discontinuing study treatment due to an AE was assessed. An AE is any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the use of the investigational product, whether or not considered related to the investigational product.
Time Frame: Up to Day 84
Population: Includes all randomized participants receiving ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 166 | 158
Participants | 18 | 25

4. Secondary Outcome: Least Squares Mean Change From Baseline in Young-Mania Rating Scale (Y-MRS) Score at Day 42
Description: The least squares mean change from baseline in Y-MRS score at day 42 was assessed. The Y-MRS is a clinician-rated instrument used for assessing the symptoms of mania, composed of 11 items. For the 11 items, scores range from 0 (symptoms absent) to, depending on the item, either 4 (7 items) or 8 (4 items). Scores for individual items add to a total score (range: 0-60), with higher scores indicating greater symptom severity. Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 42
Population: Includes all randomized participants receiving ≥1 dose of study treatment, having ≥1 post-dose Y-MRS assessment.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline | 28.2 (0.45) | 27.9 (0.46)
  Change from Baseline at Day 42 | -8.7 (0.84) | -11.4 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 42; Test type: Superiority; p = 0.0210, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

5. Secondary Outcome: Least Squares Mean Change From Baseline in Young-Mania Rating Scale (Y-MRS) Score at Day 84
Description: The least squares mean change from baseline in Y-MRS score at day 84 was assessed. The Y-MRS is a clinician-rated instrument used for assessing the symptoms of mania, composed of 11 items. For the 11 items, scores range from 0 (symptoms absent) to, depending on the item, either 4 (7 items) or 8 (4 items). Scores for individual items add to a total score (range: 0-60), with higher scores indicating greater symptom severity. Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: Includes all randomized participants receiving ≥1 dose of study treatment, having ≥1 post-dose Y-MRS assessment.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline | 28.2 (0.45) | 27.9 (0.46)
  Change from Baseline at Day 84 | -9.3 (0.89) | -12.7 (0.92)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.0073, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

6. Secondary Outcome: Number of Participants Achieving Young-Mania Rating Scale (Y-MRS) Responder Status
Description: The Y-MRS is a clinician-rated instrument used for assessing the symptoms of mania, composed of 11 items. For the 11 items, scores range from 0 (symptoms absent) to, depending on the item, either 4 (7 items) or 8 (4 items). Scores for individual items add to a total score (range: 0-60), with higher scores indicating greater symptom severity. At pre-specified time points, the number of participants achieving Y-MRS responder status was assessed, defined as the number of participants with a 50% decrease from baseline in Y-MRS total score. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Up to Day 84
Population: Includes all randomized participants receiving ≥1 dose of study treatment, having ≥1 post-dose Y-MRS assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Participants
  Day 3: number analyzed (Participants) | 154 | 142
  Day 3 | 10 | 13
  Day 7: number analyzed (Participants) | 163 | 154
  Day 7 | 25 | 22
  Day 14 | 34 | 46
  Day 21 | 44 | 53
  Day 42 | 52 | 67
  Day 63 | 52 | 66
  Day 84 | 56 | 74
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Day 3; Test type: Superiority; p = 0.3928, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 2: Comparison: Placebo vs Asenapine; Day 7; Test type: Superiority; p = 0.7923, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 3: Comparison: Placebo vs Asenapine; Day 14; Test type: Superiority; p = 0.0701, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 4: Comparison: Placebo vs Asenapine; Day 21; Test type: Superiority; p = 0.1634, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 5: Comparison: Placebo vs Asenapine; Day 42; Test type: Superiority; p = 0.0370, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 6: Comparison: Placebo vs Asenapine; Day 63; Test type: Superiority; p = 0.0488, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 7: Comparison: Placebo vs Asenapine; Day 84; Test type: Superiority; p = 0.0152, Chi-squared; Based on Pearson's chi-squared test

7. Secondary Outcome: Number of Participants Achieving Young-Mania Rating Scale (Y-MRS) Remitter Status
Description: The Y-MRS is a clinician-rated instrument used for assessing the symptoms of mania, composed of 11 items. For the 11 items, scores range from 0 (symptoms absent) to, depending on the item, either 4 (7 items) or 8 (4 items). Scores for individual items add to a total score (range: 0-60), with higher scores indicating greater symptom severity. At pre-specified time points, the number of participants achieving Y-MRS remitter status was assessed, defined as the number of participants with a Y-MRS total score of 12 or lower. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Up to Day 84
Population: Includes all randomized participants receiving ≥1 dose of study treatment, having ≥1 post-dose Y-MRS assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Participants
  Day 3: number analyzed (Participants) | 154 | 142
  Day 3 | 8 | 11
  Day 7: number analyzed (Participants) | 163 | 154
  Day 7 | 21 | 19
  Day 14 | 32 | 42
  Day 21 | 35 | 52
  Day 42 | 46 | 64
  Day 63 | 46 | 63
  Day 84 | 49 | 67
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Day 3; Test type: Superiority; p = 0.3709, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 2: Comparison: Placebo vs Asenapine; Day 7; Test type: Superiority; p = 0.8837, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 3: Comparison: Placebo vs Asenapine; Day 14; Test type: Superiority; p = 0.1153, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 4: Comparison: Placebo vs Asenapine; Day 21; Test type: Superiority; p = 0.0158, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 5: Comparison: Placebo vs Asenapine; Day 42; Test type: Superiority; p = 0.0143, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 6: Comparison: Placebo vs Asenapine; Day 63; Test type: Superiority; p = 0.0196, Chi-squared; Based on Pearson's chi-squared test
Statistical Analysis 7: Comparison: Placebo vs Asenapine; Day 84; Test type: Superiority; p = 0.0148, Chi-squared; Based on Pearson's chi-squared test

8. Secondary Outcome: Least Squares Mean Change From Baseline in Clinical Global Impressions for Use in Bipolar Disorder (CGI-BP) Severity of Mania Score at Day 21
Description: The least squares mean change from baseline in CGI-BP severity of mania score at day 21 was assessed. The CGI-BP severity of mania scale is a clinician-rated scale for assessing the severity of manic symptoms of bipolar disorder, with scores ranging from 1 (normal) to 7 (very severely ill). Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: Per protocol, the overall analysis population includes all randomized participants receiving ≥1 dose of study treatment, with ≥1 post-dose Y-MRS assessment. For Baseline / Change from Baseline data, includes only participants of the overall analysis population with an observation at the time indicated for the respective endpoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 4.5 (0.06) | 4.5 (0.07)
  Change from Baseline at Day 21: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 21 | -0.8 (0.09) | -1.1 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.0046, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

9. Secondary Outcome: Least Squares Mean Change From Baseline in Clinical Global Impressions for Use in Bipolar Disorder (CGI-BP) Severity of Mania Score at Day 84
Description: The least squares mean change from baseline in CGI-BP severity of mania score at day 84 was assessed. The CGI-BP severity of mania scale is a clinician-rated scale for assessing the severity of manic symptoms of bipolar disorder, with scores ranging from 1 (normal) to 7 (very severely ill). Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 4.5 (0.06) | 4.5 (0.07)
  Change from Baseline at Day 84: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 84 | -1.0 (0.11) | -1.5 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.0006, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

10. Secondary Outcome: Least Squares Mean Change From Baseline in Clinical Global Impressions for Use in Bipolar Disorder (CGI-BP) Severity of Depression Score at Day 21
Description: The least squares mean change from baseline in CGI-BP severity of depression score at day 21 was assessed. The CGI-BP severity of depression scale is a clinician-rated scale for assessing the severity of depressive symptoms of bipolar disorder, with scores ranging from 1 (normal) to 7 (very severely ill). Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 2.3 (0.08) | 2.3 (0.08)
  Change from Baseline at Day 21: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 21 | -0.1 (0.07) | -0.2 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.3497, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

11. Secondary Outcome: Least Squares Mean Change From Baseline in Clinical Global Impressions for Use in Bipolar Disorder (CGI-BP) Severity of Depression Score at Day 84
Description: The least squares mean change from baseline in CGI-BP severity of depression score at day 84 was assessed. The CGI-BP severity of depression scale is a clinician-rated scale for assessing the severity of depressive symptoms of bipolar disorder, with scores ranging from 1 (normal) to 7 (very severely ill). Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 2.3 (0.08) | 2.3 (0.08)
  Change from Baseline at Day 84: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 84 | -0.1 (0.09) | -0.1 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.7753, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

12. Secondary Outcome: Least Squares Mean Change From Baseline in Clinical Global Impressions for Use in Bipolar Disorder (CGI-BP) Severity of Overall Bipolar Illness Score at Day 21
Description: The least squares mean change from baseline in CGI-BP severity of severity of overall bipolar illness score at day 21 was assessed. The CGI-BP severity of overall bipolar illness scale is a clinician-rated scale for assessing the severity of overall symptoms of bipolar disorder, with scores ranging from 1 (normal) to 7 (very severely ill). Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 4.6 (0.05) | 4.6 (0.06)
  Change from Baseline at Day 21: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 21 | -0.7 (0.09) | -1.0 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.0073, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

13. Secondary Outcome: Least Squares Mean Change From Baseline in Clinical Global Impressions for Use in Bipolar Disorder (CGI-BP) Severity of Overall Bipolar Illness Score at Day 84
Description: The least squares mean change from baseline in CGI-BP severity of severity of overall bipolar illness score at day 84 was assessed. The CGI-BP severity of overall bipolar illness scale is a clinician-rated scale for assessing the severity of overall symptoms of bipolar disorder, with scores ranging from 1 (normal) to 7 (very severely ill). Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 4.6 (0.05) | 4.6 (0.06)
  Change from Baseline at Day 84: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 84 | -0.8 (0.11) | -1.2 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.0102, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

14. Secondary Outcome: Least Squares Mean Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Score at Day 21
Description: The least squares mean change from baseline in MADRS score at day 21 was assessed. The MARDS is a clinician-rated scale for assessing the severity of symptoms of depression, composed of 10 items. For the 10 items, scores range from 0 (symptoms absent) to 6 (severe). Scores for individual items add to a total score (range: 0-60), with higher scores indicating greater severity of depression. Further, decreases in depression severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 11.4 (0.48) | 11.3 (0.50)
  Change from Baseline at Day 21: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 21 | -2.2 (0.51) | -2.9 (0.54)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.3684, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

15. Secondary Outcome: Least Squares Mean Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Score at Day 84
Description: The least squares mean change from baseline in MADRS score at day 84 was assessed. The MARDS is a clinician-rated scale for assessing the severity of symptoms of depression, composed of 10 items. For the 10 items, scores range from 0 (symptoms absent) to 6 (severe). Scores for individual items add to a total score (range: 0-60), with higher scores indicating greater severity of depression. Further, decreases in depression severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 11.4 (0.48) | 11.3 (0.50)
  Change from Baseline at Day 84: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 84 | -1.7 (0.64) | -1.6 (0.68)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.9370, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

16. Secondary Outcome: Least Squares Mean Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Score at Day 21
Description: The least squares mean change from baseline in PANSS score at day 21 was assessed. The PANSS assesses the severity of schizophrenia symptoms through a clinician-rated inventory of 30 items organized in 3 subscales: 1) positive subscale (7 items); 2) negative subscale (7 items); and 3) general psychopathology subscale (16 items). For each item, symptoms are scored from 1 (absent) to 7 (extreme) and add to a total PANSS score (range: 30-210). Higher scores reflect more severe symptoms of schizophrenia. Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 67.1 (0.95) | 65.1 (0.99)
  Change from Baseline at Day 21: number analyzed (Participants) | 157 | 145
  Change from Baseline at Day 21 | -5.4 (1.09) | -7.2 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.2492, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

17. Secondary Outcome: Least Squares Mean Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Score at Day 84
Description: The least squares mean change from baseline in PANSS score at day 84 was assessed. The PANSS assesses the severity of schizophrenia symptoms through a clinician-rated inventory of 30 items organized in 3 subscales: 1) positive subscale (7 items); 2) negative subscale (7 items); and 3) general psychopathology subscale (16 items). For each item, symptoms are scored from 1 (absent) to 7 (extreme) and add to a total PANSS score (range: 30-210). Higher scores reflect more severe symptoms of schizophrenia. Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 67.1 (0.95) | 65.1 (0.99)
  Change from Baseline at Day 84: number analyzed (Participants) | 157 | 145
  Change from Baseline at Day 84 | -6.0 (1.32) | -7.4 (1.39)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.4683, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

18. Secondary Outcome: Least Squares Mean Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Score at Day 21
Description: The least squares mean change from baseline in HAM-A score at day 21 was assessed. The HAM-A is a clinician-rated instrument for assessing anxiety symptoms, composed of 14 items. For the 14 items, scores range from 0 (not present) to 4 (severe). Scores for individual items add to a total score (range: 0-56), with higher scores indicating greater severity of anxiety. Further, decreases in anxiety severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 161 | 154
  Baseline | 9.3 (0.42) | 8.8 (0.43)
  Change from Baseline at Day 21: number analyzed (Participants) | 156 | 147
  Change from Baseline at Day 21 | -2.1 (0.39) | -2.4 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.5683, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

19. Secondary Outcome: Least Squares Mean Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Score at Day 84
Description: The least squares mean change from baseline in HAM-A score at day 84 was assessed. The HAM-A is a clinician-rated instrument for assessing anxiety symptoms, composed of 14 items. For the 14 items, scores range from 0 (not present) to 4 (severe). Scores for individual items add to a total score (range: 0-56), with higher scores indicating greater severity of anxiety. Further, decreases in anxiety severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 161 | 154
  Baseline | 9.3 (0.42) | 8.8 (0.43)
  Change from Baseline at Day 84: number analyzed (Participants) | 156 | 147
  Change from Baseline at Day 84 | -2.1 (0.44) | -2.1 (0.47)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.9693, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

20. Secondary Outcome: Least Squares Mean Change From Baseline in InterSePT Scale for Suicidal Thinking - Modified Version (ISST-Modified) Score at Day 21
Description: The least squares mean change from baseline in ISST-Modified score at day 21 was assessed. The ISST-Modified is a clinician-rated scale for rating suicidality, composed of 12 items (score range: 0-2). Scores for the 12 items add to a total ISST-Modified score (range: 0-24), with higher scores indicating increased severity of suicidal thinking. Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 0.6 (0.14) | 0.4 (0.14)
  Change from Baseline at Day 21: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 21 | -0.0 (0.12) | 0.0 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.6136, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

21. Secondary Outcome: Least Squares Mean Change From Baseline in InterSePT Scale for Suicidal Thinking - Modified Version (ISST-Modified) Score at Day 84
Description: The least squares mean change from baseline in ISST-Modified score at day 84 was assessed. The ISST-Modified is a clinician-rated scale for rating suicidality, composed of 12 items (score range: 0-2). Scores for the 12 items add to a total ISST-Modified score (range: 0-24), with higher scores indicating increased severity of suicidal thinking. Further, decreases in symptom severity over time would be reflected by negative changes from baseline. For evaluation of this endpoint, a LOCF analysis was used; baseline values are not eligible to be carried forward to missing post-baseline assessments.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 162 | 154
  Baseline | 0.6 (0.14) | 0.4 (0.14)
  Change from Baseline at Day 84: number analyzed (Participants) | 162 | 154
  Change from Baseline at Day 84 | -0.0 (0.15) | 0.3 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.1586, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

22. Secondary Outcome: Mean Change From Baseline (CFB) at Day 21 in Neurocognitive Function as Determined by Central Nervous System Vital Signs (CNS-VS) Test Battery
Description: Nine neurocognitive tests with higher scores indicating better performance:
  1. Verbal Memory test: recognize/remember/retrieve words (range 0-60)
  2. Visual Memory test: recognize/remember/retrieve geometric figures (range 0-60)
  3. Speed of Processing: recognize/process information. No min./max. score. Normative average (NA); correct answers: 65.1, avg. errors: 1.37
  4. Social Acuity/Perception of Emotions test: perceive/respond to emotional cues. Min. score: -64/Max. score: 16
  5. Reasoning: reason/respond to non-verbal, visual-abstract stimuli; scores range: -15 to 15
  6. Executive Function: recognize rules/categories/decision making. No min./max. score. NA correct answers: 55.01/avg. errors: 5.28
  7. Working Memory/Continuous Performance Task (CPT): perceive/attend to symbols. Min. score: -45/Max. score: 15
  8. Sustained Attention: direct/focus on specific stimuli: Max. score (raw score); 45; Min. score: -170
  9. Composite Memory: working+verbal+visual memory, Range 0-135.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Verbal Memory - Baseline: number analyzed (Participants) | 151 | 142
  Verbal Memory - Baseline | 43.6 (9.01) | 44.6 (8.36)
  Visual Memory - Baseline: number analyzed (Participants) | 151 | 142
  Visual Memory - Baseline | 38.0 (7.89) | 38.2 (6.51)
  Processing Speed - Baseline: number analyzed (Participants) | 152 | 143
  Processing Speed - Baseline | 34.3 (25.85) | 39.5 (14.28)
  Social Acuity - Baseline: number analyzed (Participants) | 151 | 142
  Social Acuity - Baseline | 2.8 (6.90) | 2.7 (6.67)
  Reasoning - Baseline: number analyzed (Participants) | 151 | 142
  Reasoning - Baseline | 2.1 (5.54) | 1.3 (5.07)
  Executive Functioning - Baseline: number analyzed (Participants) | 151 | 142
  Executive Functioning - Baseline | 17.6 (26.06) | 16.9 (25.59)
  Working Memory - Baseline: number analyzed (Participants) | 150 | 142
  Working Memory - Baseline | 2.9 (6.56) | 2.9 (5.72)
  Sustained Attention - Baseline: number analyzed (Participants) | 150 | 142
  Sustained Attention - Baseline | 14.0 (16.83) | 13.5 (14.64)
  Composite Memory - Baseline: number analyzed (Participants) | 150 | 142
  Composite Memory - Baseline | 81.6 (15.59) | 82.8 (13.48)
  Verbal Memory - CFB at Day 21: number analyzed (Participants) | 88 | 89
  Verbal Memory - CFB at Day 21 | -0.8 (7.66) | 0.8 (8.54)
  Visual Memory - CFB at Day 21: number analyzed (Participants) | 88 | 89
  Visual Memory - CFB at Day 21 | -0.3 (8.08) | -0.4 (7.45)
  Processing Speed - CFB at Day 21: number analyzed (Participants) | 89 | 90
  Processing Speed - CFB at Day 21 | 3.8 (16.82) | 4.2 (11.97)
  Social Acuity - CFB at Day 21: number analyzed (Participants) | 89 | 89
  Social Acuity - CFB at Day 21 | 1.0 (4.76) | 0.3 (5.46)
  Reasoning - CFB at Day 21: number analyzed (Participants) | 89 | 89
  Reasoning - CFB at Day 21 | 0.3 (4.39) | 0.7 (4.33)
  Executive Functioning - CFB at Day 21: number analyzed (Participants) | 89 | 89
  Executive Functioning - CFB at Day 21 | 4.4 (16.55) | 10.1 (18.45)
  Working Memory - CFB at Day 21: number analyzed (Participants) | 87 | 89
  Working Memory - CFB at Day 21 | 0.2 (7.16) | -0.4 (5.83)
  Sustained Attention - CFB at Day 21: number analyzed (Participants) | 87 | 89
  Sustained Attention - CFB at Day 21 | 0.3 (17.23) | -0.8 (13.91)
  Composite Memory - CFB at Day 21: number analyzed (Participants) | 87 | 89
  Composite Memory - CFB at Day 21 | -1.1 (13.65) | 0.5 (13.43)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Verbal Memory - CFB at Day 21; Test type: Superiority; p = 0.0550, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 2: Comparison: Placebo vs Asenapine; Visual Memory - CFB at Day 21; Test type: Superiority; p = 0.7469, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 3: Comparison: Placebo vs Asenapine; Processing Speed - CFB at Day 21; Test type: Superiority; p = 0.3253, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 4: Comparison: Placebo vs Asenapine; Social Acuity - CFB at Day 21; Test type: Superiority; p = 0.3885, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 5: Comparison: Placebo vs Asenapine; Reasoning - CFB at Day 21; Test type: Superiority; p = 0.5975, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 6: Comparison: Placebo vs Asenapine; Executive Functioning - CFB at Day 21; Test type: Superiority; p = 0.0690, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 7: Comparison: Placebo vs Asenapine; Working Memory - CFB at Day 21; Test type: Superiority; p = 0.7970, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 8: Comparison: Placebo vs Asenapine; Sustained Attention - CFB at Day 21; Test type: Superiority; p = 0.8339, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 9: Comparison: Placebo vs Asenapine; Composite Memory - CFB at Day 21; Test type: Superiority; p = 0.2101, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

23. Secondary Outcome: Mean Change From Baseline (CFB) at Day 84 in Neurocognitive Function as Determined by Central Nervous System Vital Signs (CNS-VS) Test Battery
Description: as for outcome 22
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Verbal Memory - Baseline: number analyzed (Participants) | 151 | 142
  Verbal Memory - Baseline | 43.6 (9.01) | 44.6 (8.36)
  Visual Memory - Baseline: number analyzed (Participants) | 151 | 142
  Visual Memory - Baseline | 38.0 (7.89) | 38.2 (6.51)
  Processing Speed - Baseline: number analyzed (Participants) | 152 | 143
  Processing Speed - Baseline | 34.3 (25.85) | 39.5 (14.28)
  Social Acuity - Baseline: number analyzed (Participants) | 151 | 142
  Social Acuity - Baseline | 2.8 (6.90) | 2.7 (6.67)
  Reasoning - Baseline: number analyzed (Participants) | 151 | 142
  Reasoning - Baseline | 2.1 (5.54) | 1.3 (5.07)
  Executive Functioning - Baseline: number analyzed (Participants) | 151 | 142
  Executive Functioning - Baseline | 17.6 (26.06) | 16.9 (25.59)
  Working Memory - Baseline: number analyzed (Participants) | 150 | 142
  Working Memory - Baseline | 2.9 (6.56) | 2.9 (5.72)
  Sustained Attention - Baseline: number analyzed (Participants) | 150 | 142
  Sustained Attention - Baseline | 14.0 (16.83) | 13.5 (14.64)
  Composite Memory - Baseline: number analyzed (Participants) | 150 | 142
  Composite Memory - Baseline | 81.6 (15.59) | 82.8 (13.48)
  Verbal Memory - CFB at Day 84: number analyzed (Participants) | 98 | 98
  Verbal Memory - CFB at Day 84 | -0.0 (7.97) | -0.3 (8.63)
  Visual Memory - CFB at Day 84: number analyzed (Participants) | 98 | 98
  Visual Memory - CFB at Day 84 | 0.0 (7.47) | -0.5 (7.19)
  Processing Speed - CFB at Day 84: number analyzed (Participants) | 98 | 99
  Processing Speed - CFB at Day 84 | 3.6 (16.31) | -1.4 (61.50)
  Social Acuity - CFB at Day 84: number analyzed (Participants) | 98 | 98
  Social Acuity - CFB at Day 84 | 0.7 (5.04) | 0.9 (5.70)
  Reasoning - CFB at Day 84: number analyzed (Participants) | 98 | 98
  Reasoning - CFB at Day 84 | -0.1 (4.81) | 1.0 (4.88)
  Executive Functioning - CFB at Day 84: number analyzed (Participants) | 98 | 98
  Executive Functioning - CFB at Day 84 | 3.9 (19.37) | 10.2 (19.97)
  Working Memory - CFB at Day 84: number analyzed (Participants) | 97 | 98
  Working Memory - CFB at Day 84 | -0.2 (7.06) | -0.4 (5.98)
  Sustained Attention - CFB at Day 84: number analyzed (Participants) | 97 | 98
  Sustained Attention - CFB at Day 84 | -0.5 (18.17) | 0.5 (15.11)
  Composite Memory - CFB at Day 84: number analyzed (Participants) | 97 | 98
  Composite Memory - CFB at Day 84 | -0.0 (14.16) | -0.7 (13.63)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Verbal Memory - CFB at Day 84; Test type: Superiority; p = 0.6914, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 2: Comparison: Placebo vs Asenapine; Visual Memory - CFB at Day 84; Test type: Superiority; p = 0.8805, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 3: Comparison: Placebo vs Asenapine; Processing Speed - CFB at Day 84; Test type: Superiority; p = 0.4878, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 4: Comparison: Placebo vs Asenapine; Social Acuity - CFB at Day 84; Test type: Superiority; p = 0.8051, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 5: Comparison: Placebo vs Asenapine; Reasoning - CFB at Day 84; Test type: Superiority; p = 0.1925, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 6: Comparison: Placebo vs Asenapine; Executive Functioning - CFB at Day 84; Test type: Superiority; p = 0.0514, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 7: Comparison: Placebo vs Asenapine; Working Memory - CFB at Day 84; Test type: Superiority; p = 0.9898, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 8: Comparison: Placebo vs Asenapine; Sustained Attention - CFB at Day 84; Test type: Superiority; p = 0.5683, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 9: Comparison: Placebo vs Asenapine; Composite Memory - CFB at Day 84; Test type: Superiority; p = 0.8907, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

24. Secondary Outcome: Percentage of Participants Determined to be Ready to Discharge at Day 84 (Kaplan-Meier Estimation)
Description: The percentage of participants determined to be ready to discharge at day 84 was estimated (Kaplan-Meier), using the readiness to discharge questionnaire (RDQ). The RDQ is clinician-rated scale to assess readiness for discharge, composed of 7 items. Of the 7 items, only the first 5 items were utilized:
  1. Not actively suicidal/homicidal;
  2. Adequate control over aggression and impulsivity;
  3. Able to carry out basic activities of daily life;
  4. Able to take medicine independently; and
  5. Delusions and hallucinations do not significantly interfere with functioning.
  For the 5 items, the clinician provided a response (Strongly Disagree; Disagree; Agree; or Strongly Agree) at each pre-specified visit. The first visit at which the responses to the first 5 items on the RDQ are "Strongly Agree" or "Agree," was defined as the point a participant was ready to discharge.
Time Frame: Day 84
Population: Per protocol, the analysis population for this endpoint includes all randomized participants receiving ≥1 dose of study treatment, with ≥1 post-dose Y-MRS assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Percentage of Participants | 74.1 [64.0 to 84.2] | 89.7 [75.0 to 100.0]
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Test type: Superiority; p = 0.0613, Log Rank

25. Secondary Outcome: Least Squares Mean Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q), General Activities Subscale Score at Day 21
Description: The least squares mean change from baseline in Q-LES-Q score at day 21 was assessed. The Q-LES-Q is a participant-completed questionnaire to assess general satisfaction with activities such as physical health, mood, work, household tasks, social and family relationships, leisure activities, and overall satisfaction, composed of 16 items. For each of the 16 items, scores range from 0 (very poor) to 5 (very good), with scores for all items adding to a total score (range: 0-80); higher scores indicate better quality of life. Further, decreases in quality of life are reflected by a negative change from baseline.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 155 | 148
  Baseline | 61.0 (1.53) | 61.3 (1.58)
  Change from Baseline at Day 21: number analyzed (Participants) | 88 | 91
  Change from Baseline at Day 21 | 3.9 (1.63) | 4.6 (1.50)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 21; Test type: Superiority; p = 0.7493, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

26. Secondary Outcome: Least Squares Mean Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q), General Activities Subscale Score at Day 84
Description: The least squares mean change from baseline in Q-LES-Q score at day 84 was assessed. The Q-LES-Q is a participant-completed questionnaire to assess general satisfaction with activities such as physical health, mood, work, household tasks, social and family relationships, leisure activities, and overall satisfaction, composed of 16 items. For each of the 16 items, scores range from 0 (very poor) to 5 (very good), with scores for all items adding to a total score (range: 0-80); higher scores indicate better quality of life. Further, decreases in quality of life are reflected by a negative change from baseline.
Time Frame: Baseline and Day 84
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  Baseline: number analyzed (Participants) | 155 | 148
  Baseline | 61.0 (1.53) | 61.3 (1.58)
  Change from Baseline at Day 84: number analyzed (Participants) | 41 | 46
  Change from Baseline at Day 84 | -3.7 (3.10) | -1.1 (2.60)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; Change from Baseline at Day 84; Test type: Superiority; p = 0.4884, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

27. Secondary Outcome: Least Squares Mean Change From Baseline at Day 21 in Quality of Life as Determined by Short Form-36 Version 2 (SF-36v2)
Description: Least squares mean change from baseline at day 21 in quality of life was assessed, as determined by SF-36v2. The SF-36v2 is a self-administered questionnaire, measuring 8 domains: Physical Functioning (PF); Role-Physical (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role-Emotional (RE); and Mental Health (MH). These 8 concepts are further organized into a Physical Component Summary (PCS; composite of PF, RP, BP, and GH) and a Mental Component Summary (MCS; composite of VT, SF, RE, and MH). The SF-36v2 domains and composite summaries were scored using a norm-based scoring approach, yielding a mean of 50 and standard deviation of 10 based on the norms from the 1998 SF-36 United States general population norms. For the PCS and MCS, scores range from 0 to 100, with higher scores indicating better quality of life. Further, decreases in quality of life (by PCS and MCS) are reflected by a negative change from baseline.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  PCS - Baseline: number analyzed (Participants) | 153 | 148
  PCS - Baseline | 50.49 (0.728) | 51.64 (0.739)
  PCS - Change from Baseline at Day 21: number analyzed (Participants) | 88 | 91
  PCS - Change from Baseline at Day 21 | -0.72 (0.929) | -2.47 (0.848)
  MCS - Baseline: number analyzed (Participants) | 153 | 148
  MCS - Baseline | 40.83 (1.085) | 39.03 (1.100)
  MCS - Change from Baseline at Day 21: number analyzed (Participants) | 88 | 91
  MCS - Change from Baseline at Day 21 | 2.29 (1.273) | 5.93 (1.174)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; PCS - Change from Baseline at Day 21; Test type: Superiority; p = 0.1280, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 2: Comparison: Placebo vs Asenapine; MCS - Change from Baseline at Day 21; Test type: Superiority; p = 0.0215, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

28. Secondary Outcome: Least Squares Mean Change From Baseline at Day 84 in Quality of Life as Determined by Short Form-36 Version 2 (SF-36v2)
Description: Least squares mean change from baseline at day 84 in quality of life was assessed, as determined by SF-36v2. The SF-36v2 is a self-administered questionnaire, measuring 8 domains: Physical Functioning (PF); Role-Physical (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role-Emotional (RE); and Mental Health (MH). These 8 concepts are further organized into a Physical Component Summary (PCS; composite of PF, RP, BP, and GH) and a Mental Component Summary (MCS; composite of VT, SF, RE, and MH). The SF-36v2 domains and composite summaries were scored using a norm-based scoring approach, yielding a mean of 50 and standard deviation of 10 based on the norms from the 1998 SF-36 United States general population norms. For the PCS and MCS, scores range from 0 to 100, with higher scores indicating better quality of life. Further, decreases in quality of life (by PCS and MCS) are reflected by a negative change from baseline.
Time Frame: Baseline and Day 21
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Asenapine
Number analyzed (Participants) | 163 | 155
Score on a Scale
  PCS - Baseline: number analyzed (Participants) | 153 | 148
  PCS - Baseline | 50.49 (0.728) | 51.64 (0.739)
  PCS - Change from Baseline at Day 84: number analyzed (Participants) | 42 | 46
  PCS - Change from Baseline at Day 84 | 1.37 (1.238) | -0.95 (1.079)
  MCS - Baseline: number analyzed (Participants) | 153 | 148
  MCS - Baseline | 40.83 (1.085) | 39.03 (1.100)
  MCS - Change from Baseline at Day 84: number analyzed (Participants) | 42 | 46
  MCS - Change from Baseline at Day 84 | -1.05 (2.278) | 2.49 (1.985)
Statistical Analysis 1: Comparison: Placebo vs Asenapine; PCS - Change from Baseline at Day 84; Test type: Superiority; p = 0.1331, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate
Statistical Analysis 2: Comparison: Placebo vs Asenapine; MCS - Change from Baseline at Day 84; Test type: Superiority; p = 0.2024, ANCOVA — P-value based on the difference in the LS means for asenapine versus placebo; Based on an ANCOVA model with treatment and pooled investigative site as fixed effects and baseline as a covariate

ADVERSE EVENTS:
Time Frame: Up to Day 114
Description: Includes all participants receiving study treatment. Additionally, serious adverse events were coded using MedDRA 10, while other adverse events were coded using MedDRA 9.1.
Arm/Group | Placebo | Asenapine
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/158
Serious Adverse Events (participants affected / at risk) | 24/166 | 21/158
Other Adverse Events (participants affected / at risk) | 76/166 | 91/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=166) | Asenapine (N=158)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Arthritis Bacterial (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Malaria (Infections and infestations) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 1
Bipolar I Disorder (Psychiatric disorders) | 1 | 3
Depression (Psychiatric disorders) | 3 | 3
Depressive Symptom (Psychiatric disorders) | 0 | 2
Major Depression (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 13 | 8
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Drug Abuser (Social circumstances) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=166) | Asenapine (N=158)
Diarrhoea (Gastrointestinal disorders) | 12 | 3
Nausea (Gastrointestinal disorders) | 10 | 10
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 9
Weight Increased (Investigations) | 1 | 8
Headache (Nervous system disorders) | 23 | 22
Tremor (Nervous system disorders) | 9 | 7
Akathisia (Nervous system disorders) | 9 | 5
Sedation (Nervous system disorders) | 10 | 21
Somnolence (Nervous system disorders) | 7 | 18
Dizziness (Nervous system disorders) | 5 | 8
Agitation (Psychiatric disorders) | 9 | 10
Insomnia (Psychiatric disorders) | 16 | 20
Mania (Psychiatric disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except for compelling legal reasons, neither the sponsor nor the investigator will communicate to third parties any result of the clinical trial before the clinical trial report (CTR) has been released by the sponsor.